CLINICAL TRIAL: NCT03325764
Title: Fitness, Physical Activity and Movement Analysis in Obese Patients Undergoing Bariatric Surgery
Acronym: FAMOUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HAO 017013; 2017-A01807-46 (Other: ANSM)
Record Dates: First submitted 2017-10-12; First posted 2017-10-30 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Sleeve Gastrectomy
Keywords: Obesity; bariatric surgery; sleeve gastrectomy; physical activity; movement analysis
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Longitudinal study comparing data before bariatric surgery and one year after bariatric surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sleeve gastrectomy (Other): Assessment before and after sleeve gastrectomy
  Interventions: Other: functional assessment

INTERVENTIONS:
Other: functional assessment — assessment of functional capacity, habitual physical, cardiorespiratory fitness, muscle power and postural stability and gait parameters

SUMMARY:
This study aims to describe the effects of sleeve gastrectomy, the most commonly performed bariatric procedure worldwide, on functional capacity, habitual physical activity, physical fitness (cardiorespiratory and muscular fitness) and gait parameters in severely obese subjects undergoing bariatric surgery. Functional capacity, physical activity, physical fitness and gait parameters will be objectively assessed and compared among candidates seeking sleeve gastrectomy and 6 months after sleeve gastrectomy.

DETAILED DESCRIPTION:
This study is a monocentric longitudinal study conducting in obese patients: candidates to sleeve gastrectomy and these same patients 6 months after.The primary aim of this study is to describe the effects of sleeve gastrectomy on habitual physical activity, physical fitness (cardiorespiratory and muscular fitness) and gait parameters in severely obese patients. Functional capacity will be assessed during a 6-min walk test, habitual physical activity with accelerometers during 7-day recordings in habitual life conditions (Actigraph GT3X® and activPAL®), cardiorespiratory fitness during a maximal exercise test on a cycle ergometer with a direct measure of peakVO2, muscle strength with an isokinetic dynamometer (Contrex®), muscle power and postural stability with force platforms (Kistler® and Satel®) and gait parameters with a gait analysis system (GaitRite®). Fatigue, quality of life and joint pain will be assessed with questionnaires (MFI-20, SF36 and WOMAC, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age between 18 and 65 years
* Planned obesity treatment by sleeve gastrectomy
* Patient with massive obesity (BMI ≥ 40 kg/m2) or severe obesity (BMI between 35 and 40 kg/m2) with comorbidities
* Written informed consent

Exclusion Criteria:

* Subject not affiliated with a social security scheme
* Regular follow-up not feasible
* Participation in a structured physical activity program
* Severe orthopedic problems
* Disabling neuropathy
* Recent (< 6 months) coronary event
* Abnormal cardiac stress test
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
functional capacity | before and 6 months after sleeve gastrectomy
  Difference in functional capacity (6-min walk test distance)

SECONDARY OUTCOMES:
habitual physical activity (Actigraph GT3X® and activPAL®) | before and 6 months after sleeve gastrectomy
  Difference in habitual physical activity
cardiorespiratory fitness ( cycle ergometer ) | before and 6 months after sleeve gastrectomy
  Difference in cardiorespiratory fitness
muscle strength ( isokinetic dynamometer (Contrex®)) | before and 6 months after sleeve gastrectomy
  Difference in muscle strength

CONTACTS AND LOCATIONS:
Locations (1):
- GH-Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bellicha A, Giroux C, Ciangura C, Menoux D, Thoumie P, Oppert JM, Portero P. Vertical Jump on a Force Plate for Assessing Muscle Strength and Power in Women With Severe Obesity: Reliability, Validity, and Relations With Body Composition. J Strength Cond Res. 2022 Jan 1;36(1):75-81. doi: 10.1519/JSC.0000000000003432. PMID 32218061